CLINICAL TRIAL: NCT04696276
Title: Implementing Enhanced Recovery After Surgery (ERAS) Pathways In Major Gynecologic Oncology Operations In Greece
Acronym: ERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, MARIA BOURAZANI, Registered Nurse, PhD candidate, Saint Savvas Anticancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 8/11-09-2019
Record Dates: First submitted 2020-11-08; First posted 2021-01-06 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer; Hysterectomy; Endometrial Cancer; Gynecologic Cancer
Keywords: gynecologic cancer; ERAS protocols; ERAS pathways; Gynecologic/oncology surgery
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-ERAS (Experimental): will receive ERAS pathways care
  Interventions: Other: ERAS protocol
- B-nonERAS (No Intervention): will receive traditional non ERAS care

INTERVENTIONS:
Other: ERAS protocol — special approaches in three phases preoperatively, intraoperatively and postoperatively, by an interdisciplinary team comprising of the surgeon, the anesthesiologist and the nurse. The combination of these techniques reduces the reaction to postoperative stress, relieves acute postoperative pain, restores the patient immediately to their original feeding and mobilization habits, thus reducing the time required for their complete recovery.
  Arms: A-ERAS

SUMMARY:
The Enhanced Recovery After Surgery (ERAS) program includes preoperative counseling, fasting avoidance, non-opioid analgesia, fluid balance, normothermia and early mobilization. ERAS pathways were developed to reduce hospital length of stay, reduce costs and decrease perioperative opioid requirements, and be beneficial for patients. We propose the hypothesis that the ERAS pathway could reduce the length of stay (LOS) in hospital for patients undergoing major gynecologic oncology surgery (MGOS).

Patients were randomly allocated in two groups: An ERAS pathway group including preoperative counseling, early feeding/mobilization, and opioid-sparing multimodal analgesia; and a classic model group of post operative recovery as control.

DETAILED DESCRIPTION:
The Gynecological Cancer of the inner genital organs includes ovarian cancer, endometrial and cervical cancer and its therapeutic approach is surgical removal of the organ with cancer.

The last decade has developed various postoperative recovery protocols aimed at safe and rapid recovery of the patient after a surgery and early discharge from the hospital. These protocols are known as ERAS (Enhanced Recovery After Surgery) protocols or Fast-Track (FT) and combine various evidence-based perioperative care techniques.

The ERAS protocols include specific approaches preoperative, intraoperative and postoperative, by the multidisciplinary team (surgeon, anesthetist and nurse), and aim at reducing the postoperative stress and pain, fasten the feeding and the mobilization of the patient after the surgery and rapid the hospital discharge.

This trial is designed to evaluate the superiority of the ERAS pathway to conventional non-ERAS clinical practice in reducing the LOS. The results may provide new insight into the clinical applications of the ERAS pathway for MGOS.

This doctoral thesis aims to compare the effectiveness of the Protocol ERAS against the classical model of recovery, in the postoperative recovery of patients with Gynecological Cancer undergoing MGOS, in a Public Oncology Hospital in Greece.

The importance of ERAS programs is expected to emerge in the length of hospital stay, in pain control, in perioperative stress, in the early feeding and mobilization of patients who have undergone MGOS.

ELIGIBILITY:
Inclusion Criteria:

* Greek language speakers
* Have complete mental clarity
* Age >18 years

Exclusion Criteria:

* Refusal to sign consent
* Patients receiving treatment for chronic pain
* Patients receiving antipsychotic therapy, Psychopathy
* They have acute or chronic kidney and / or liver disease
* History or family history of malignant hyperthermia
* Known allergy to propofol, desflurane, or any other anesthetic agent
* Impairment of cognitive function or communication
* History of postoperative delirium

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MARIA BOURAZANI, PhD, Principal Investigator — Saint Savvas Anticancer Hospital
Locations (1):
- Saint Savvas Anticancer Hospital, Athens, Attica, Greece

REFERENCES:
- See also: Original Paper — https://www.vima-asklipiou.gr/en/articles/Protokollo-taxeias-metegxeirhtikhs-anarroshs-se-meizones-ogkologikes-gunaikologikes-epemvaseis/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between January 2020 and December 2021 from a General Anticancer Oncology Centre of Athens, Greece.
Pre-assignment Details: After obtaining consent, participants were screened for for study inclusion criteria. If entry criteria were passed they were randomized to the study.
Groups:
- A-ERAS: N=51 following the ERAS protocol
- B-Non ERAS: N=50 following a conventional post-op care
Period: Overall Study
Arm/Group | A-ERAS | B-Non ERAS
Started | 51 | 50
Completed | 51 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- A-ERAS: following the ERAS protocol
- B-Non ERAS: following a conventional post-op care
- Total: Total of all reporting groups
Arm/Group | A-ERAS | B-Non ERAS | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 34 | 77
  >=65 years | 8 | 16 | 24
Sex: Female, Male [Count of Participants; unit: Participants] — Participants were only female
  Participants
    Female | 51 | 50 | 101
    Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.4 (0.7) | 26.8 (0.7) | 26.6 (0.7)
Marital status [Count of Participants; unit: Participants]
  unmarried | 13 | 5 | 18
  married | 23 | 32 | 55
  divorced | 10 | 7 | 17
  widowed | 5 | 6 | 11
Number of Children [Count of Participants; unit: Participants]
  No children | 14 | 5 | 19
  1 child | 4 | 7 | 11
  2 children | 20 | 25 | 45
  >2 children | 13 | 13 | 26
educational level [Count of Participants; unit: Participants]
  primary school | 7 | 7 | 14
  high school | 18 | 25 | 43
  college / university | 19 | 11 | 30
  MSc / PhD | 7 | 7 | 14
Profession [Count of Participants; unit: Participants]
  housewives / students | 5 | 6 | 11
  unemployed | 4 | 8 | 12
  workers | 31 | 24 | 55
  pensioners | 11 | 12 | 23
Smoking [Count of Participants; unit: Participants]
  smokers | 18 | 22 | 40
  non-smokers | 33 | 28 | 61
alcohol consumption [Count of Participants; unit: Participants]
  0-1 drink per week | 45 | 41 | 86
  2+ drinks per week | 6 | 9 | 15
endocrinological diseases [Count of Participants; unit: Participants]
  yes | 20 | 21 | 41
  none | 31 | 29 | 60
Urinary tract diseases [Count of Participants; unit: Participants]
  yes | 0 | 2 | 2
  none | 51 | 48 | 99
kidney or liver disease [Count of Participants; unit: Participants]
  yes | 3 | 6 | 9
  none | 48 | 44 | 92
Cardiovascular diseases [Count of Participants; unit: Participants]
  yes | 12 | 15 | 27
  none | 39 | 35 | 74
Diseases of the respiratory system [Count of Participants; unit: Participants]
  yes | 6 | 5 | 11
  none | 45 | 45 | 90
Diseases of the digestive system [Count of Participants; unit: Participants]
  yes | 5 | 3 | 8
  none | 46 | 47 | 93
nervous system diseases [Count of Participants; unit: Participants]
  yes | 5 | 4 | 9
  none | 46 | 46 | 92
Skin diseases [Count of Participants; unit: Participants]
  yes | 1 | 1 | 2
  no | 50 | 49 | 99
other malignancy [Count of Participants; unit: Participants]
  had other cancer in the past | 13 | 6 | 19
  had not cancer in the past | 38 | 44 | 82
Allergies [Count of Participants; unit: Participants]
  yes | 12 | 9 | 21
  no | 39 | 41 | 80
Hemoglobin [Mean (Standard Deviation); unit: g/dl] | 12.7 (1.1) | 12.6 (1.5) | 12.65 (1.3)
Hematocrit [Mean (Standard Deviation); unit: percentage % of red blood cells in blood] | 38.9 (3.2) | 38.7 (4.5) | 38.8 (3.85)
WBC [Mean (Standard Deviation); unit: g/dl] | 6.9 (2) | 7.6 (2.1) | 7.25 (2.05)
Glucose [Mean (Standard Deviation); unit: mg/dl] | 96.7 (20.9) | 101 (21.2) | 98.85 (21.05)
Plasma proteins [Mean (Standard Deviation); unit: g/dl] | 7.1 (0.6) | 7.2 (0.6) | 7.15 (0.6)
Albumin [Mean (Standard Deviation); unit: g/dl] | 4.2 (0.4) | 4.3 (0.5) | 4.25 (0.45)

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay (LOS)
Description: Measuring how many days the participants will stay in hospital for the post-op recovery. It is defined as the time frame from the day of the surgery to the day of discharge from the hospital (unit: days).
Time Frame: up to 30 postoperative days
Measure: Mean (Inter-Quartile Range); unit: days
Groups:
- LOS in ERAS Group: Participants in ERAS group had received the enhanced recovery after surgery care
- LOS in Non-ERAS Group: Participants in the non-ERAS group had received the convectional care after surgery
Arm/Group | LOS in ERAS Group | LOS in Non-ERAS Group
Number analyzed (Participants) | 51 | 50
days | 3.8 [2 to 10] | 5.9 [3 to 10]

2. Primary Outcome: Pain Levels
Description: Evaluation of analgesia and correlation of requirements with opioid analgesics; by recording of postoperative pain levels and the evaluation of the effectiveness of analgesic treatment of patients. Using Numbered pain Scale, from 0 that means no pain at all, to 10 that means the worst pain.
  As lower the number on pain scale as better the outcome.
Time Frame: up to 3 postoperative days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Postoperative Pain Levels in ERAS Group: The ERAS group had IV parecoxib 40mg, acetaminophen (paracetamol) 1gr, morfine 0.1mg/kg and MgSO4 25% intraoperatively and postoperatively on the same day (Day-0).
  From the Day-1 until the dischard the ERAS group had PO tb oxycodone 5mg/paracetamol 325mg q:4-6 prn and lornoxicam 8mg x 2
- Postoperative Pain Levels in Non-ERAS Group: The non-ERAS group had IV parecoxib 40mg, paracetamol 1gr and Morfine 0.1mg/kg intraoperatively and paracetamol 1gr x4, tramadol 50-100mg x4, postoperatively from Day-0 until the Day-3. From the Day-4 until the dischard the non-ERAS group had PO tb paracetamol 400mg /codeine10mg/cafeine 50mg X3.
Arm/Group | Postoperative Pain Levels in ERAS Group | Postoperative Pain Levels in Non-ERAS Group
Number analyzed (Participants) | 51 | 50
units on a scale | 3.6 (1) | 4.6 (1.2)

3. Primary Outcome: Number of Participants With the Ability to Getting up in a Chair Within 18h
Description: The number of participants who had the ability to have a sit steadily on a chair himself, within the first 18 hours after the surgery.
Time Frame: within the first 18 postoperative hours
Measure: Count of Participants; unit: Participants
Groups:
- Sitting -up on a Chair for Participants in ERAS Group: Participants in ERAS group were sat on a chair within the first 18 postoperative hours
- Sitting-up on a Chair for Participants in Non-ERAS Group: Participants in non-ERAS group were sat on a chair within the first 18 postoperative hours
Arm/Group | Sitting -up on a Chair for Participants in ERAS Group | Sitting-up on a Chair for Participants in Non-ERAS Group
Number analyzed (Participants) | 49 | 49
Participants | 46 | 5

4. Primary Outcome: Number of Participants With the Ability of Full Mobilization Within 18h Postoperatively
Description: The participants should be able to stand on their feet, walk in the room, go to the toilet and make a short walk in the surgical ward within the first 18 hours after the surgery.
  Mobilization time, which is defined as the time frame from the end of the operation until they are able to walk without external assistance (unit: hours).
Time Frame: within the first 18 hours after the surgery
Measure: Count of Participants; unit: Participants
Groups:
- Standing-up in the Room for Participants in ERAS Group: Participants in ERAS group were stand-up in the first 18 postoperative hours
- Standing-up in the Room for Participants in Non-ERAS Group: Participants in non-ERAS group were stand-up for the first 18 postoperative hours
Arm/Group | Standing-up in the Room for Participants in ERAS Group | Standing-up in the Room for Participants in Non-ERAS Group
Number analyzed (Participants) | 50 | 49
Participants | 48 | 9

5. Primary Outcome: Early Feeding
Description: Feeding within the first 6 hours after the surgery. The participants should be able to drink clear fluids (water, tea,chamomile, apple juice, filter coffee, jelo) with or without sweeteners, given that they don't have PONV.
Time Frame: up to 6 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | A-ERAS | B-Non ERAS
Number analyzed (Participants) | 50 | 49
Participants | 44 | 2

6. Secondary Outcome: Early Mobilization of the Digestive System
Description: Number of participants who had their digestive system function on time, with hunger, bowel sounds and bowel movements within the first 24 hours postoperatively
Time Frame: within 24 hours post surgery
Measure: Count of Participants; unit: Participants
Groups:
- A-ERAS: The functionality of the digestive tract was assessed and if deemed necessary the patient received mild laxatives.
- B-Non ERAS: Following a conventional post-op care. Bowel function testing
Arm/Group | A-ERAS | B-Non ERAS
Number analyzed (Participants) | 50 | 49
Participants | 46 | 8

7. Secondary Outcome: Early Discontinuation of IV Administration
Description: Number of participants who had early discontinuation of IV fluids and conversion to per os within 24 hours postoperatively
Time Frame: within 24 h post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | A-ERAS | B-Non ERAS
Number analyzed (Participants) | 50 | 49
Participants | 41 | 2

8. Secondary Outcome: Number of Participants Who Had Their Urinary Catheter Removal
Description: Number of participants who had their urinary catheter removed within 24 hours postoperatively
Time Frame: within the first 24h after surgery
Measure: Count of Participants; unit: Participants
Groups:
- ERAS Group Urinary Catheter Removal: Participants in ERAS group were the urinary catheter removed within 24hour post surgery
- Non-ERAS Group Urinary Catheter Removal: Participants in non-ERAS group were the urinary catheter removed within 24h post surgery
Arm/Group | ERAS Group Urinary Catheter Removal | Non-ERAS Group Urinary Catheter Removal
Number analyzed (Participants) | 45 | 44
Participants | 43 | 6

9. Secondary Outcome: Number of Participants Who Had Their Drainage Removal Within 24h
Description: Number of Participants who had their drainage removal within 24 hours postoperatively
Time Frame: within 24h post surgery
Measure: Count of Participants; unit: Participants
Groups:
- A-ERAS Group: following the ERAS protocol.
- B-Non ERAS Group: following a conventional post-op care
Arm/Group | A-ERAS Group | B-Non ERAS Group
Number analyzed (Participants) | 50 | 49
Participants | 48 | 16

10. Secondary Outcome: Blood Transfusion
Description: Number of participants who had blood transfusion during their intraoperative and postoperative time
Time Frame: within 48 hours post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | A-ERAS | B-Non ERAS
Number analyzed (Participants) | 51 | 50
Participants | 0 | 9

11. Secondary Outcome: Postoperative Complications
Description: The evaluation of postoperative complications such as bleeding, thrombosis and inflammation.
Time Frame: up to 5 postoperative days
Measure: Number; unit: participants
Groups:
- Complication in ERAS Group: Number of participants were had post-op complication following ERAS protocol
- Complications in Non-ERAS Group: Number of participants were had post-op complication following the convectional post-op care
Arm/Group | Complication in ERAS Group | Complications in Non-ERAS Group
Number analyzed (Participants) | 50 | 49
participants
  nausea | 16 | 22
  vomiting | 9 | 18
  somnolence | 4 | 17
  repression | 2 | 10
  bleeding | 1 | 5
  fever | 1 | 11
  urinary tract infection | 0 | 4
  re-operation | 1 | 2
  postoperative bilirubin | 11 | 16

12. Secondary Outcome: Readmission
Description: Readmission rate by 30 days after discharge from the hospital
Time Frame: up to 30 postoperative days
Measure: Number; unit: participants
Groups:
- ERAS Group: Participants in ERAS group had received the enhanced recovery after surgery care
- Non-ERAS Group: Participants in non-ERAS group had received the convectional post-op care
Arm/Group | ERAS Group | Non-ERAS Group
Number analyzed (Participants) | 51 | 50
participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Initial 30 postoperative days following surgical intevention
Groups:
- Number of Adverse Events in ERAS Group: Number of adverse events in participants following the ERAS protocol
- Number of Adverse Events in Non-ERAS Group: Number of adverse events in participants following the convectional post-op care
Arm/Group | Number of Adverse Events in ERAS Group | Number of Adverse Events in Non-ERAS Group
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 0/51 | 0/50

LIMITATIONS AND CAVEATS:
The limitations of the study could be the sample size (101 participants), but due to the COVID-19 pandemic where the annual number of surgeries was necessarily reduced, this number of participants is completely satisfactory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT04696276/Prot_SAP_ICF_001.pdf